CLINICAL TRIAL: NCT00923221
Title: Collection of Blood From Patients With Prostate Cancer
Status: Recruiting | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 070100; 07-C-0100; NCT00899249 (obsolete NCT alias)
Record Dates: First submitted 2009-06-17; First posted 2009-06-18 (Estimated); Last update posted 2026-01-22 (Actual); Status verified 2026-01-20

CONDITIONS: Cancer Of Prostate; Prostate Cancer; Prostatic Neoplasms; Metastatic Prostate Cancer; Prostate
Keywords: Genetic; Prostatic Neoplasms; Genotyping; Venipuncture; Polymorphism; Natural History; Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1/Participant samples: Blood samples from participants with diagnosed prostate cancer

SUMMARY:
Background:

* It is not fully understood why prostate cancer in some men becomes androgen-independent (no longer responds to anti-androgen medication), but genetics likely plays an important role.
* Genes contain the hereditary information that is passed down from parents to children. Although everyone has the same set of genes, individuals can have different forms of the same gene.
* Differences in genes may explain, at least in part, why some people develop a more aggressive form of prostate cancer than others.

Objectives:

-To obtain blood samples from patients with prostate cancer to try to identify gene differences associated with progression to the androgen independent state.

Eligibility:

-All participants participating in NCI prostate cancer protocols.

Design:

* Participants with prostate cancer are evaluated in the NCI s Medical Oncology Clinic.
* Blood samples are collected at the initial visit or at follow-up visits.
* DNA (genetic material) and white blood cells are extracted from these samples to be used for genotyping and establishment of cell lines.
* Gene variations are correlated with prostate cancer prognosis and prognostic indicators.

DETAILED DESCRIPTION:
Objectives:

-To obtain blood samples from patients with prostate cancer for genotyping analyses.

Eligibility:

- All patients seen in the NCI prostate cancer clinic are eligible.

Design:

* Patients with a prior diagnosis of prostate cancer will be evaluated in the GMB Clinic, NCI.
* Blood samples will be collected after the participant signs the protocol consent form. In general, blood will be collected for genomic DNA one time for this study. Extra samples may be requested if the original sample was not enough. The additional sample can range from one to two tubes of blood (approximately 2-3 teaspoons total). Genomic DNA and white blood cells will each be extracted from these samples to be utilized for genotyping and establishment of individual cell lines.
* Genetic variance will be correlated with prostate cancer prognosis (i.e. time from diagnosis to death) and prognostic indicators (i.e. histological tumor grade).
* Blood samples for the extraction of cell-free DNA (cfDNA) and cell-free RNA (cfRNA) may be collected at multiple timepoints for future investigations
* Healthy controls will not be compared and no correlations will be made with prostate cancer susceptibility.

ELIGIBILITY:
* INCLUSION CRITERIA:

Individuals 18 years of age and older are eligible.

Individuals with a diagnosis of prostate cancer are eligible.

EXCLUSION CRITERIA:

Children are not eligible.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary clinical
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2007-02-28 (Actual)

PRIMARY OUTCOMES:
Acquisition and longitudinal analysis of genomic DNA, cfDNA, and cfRNA from participants with prostate cancer | study duration
  Acquisition and longitudinal analysis of genomic DNA, cfDNA, and cfRNA from participants with prostate cancer to aid in understanding the mechanisms of prostate carcinogenesis and progression

CONTACTS AND LOCATIONS:
Overall Officials: William D Figg, Pharm.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request. @@@@@@In addition, all large scale genomic sequencing data will be shared with subscribers to dbGaP.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.@@@@@@Genomic data are available once genomic data are uploaded per protocol GDS plan for as long as database is active.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI.@@@@@@Genomic data are made available via dbGaP through requests to the data custodians.

REFERENCES:
- [Background] Eisenberger MA, Blumenstein BA, Crawford ED, Miller G, McLeod DG, Loehrer PJ, Wilding G, Sears K, Culkin DJ, Thompson IM Jr, Bueschen AJ, Lowe BA. Bilateral orchiectomy with or without flutamide for metastatic prostate cancer. N Engl J Med. 1998 Oct 8;339(15):1036-42. doi: 10.1056/NEJM199810083391504. PMID 9761805
- [Background] Eisenberger MA, Simon R, O'Dwyer PJ, Wittes RE, Friedman MA. A reevaluation of nonhormonal cytotoxic chemotherapy in the treatment of prostatic carcinoma. J Clin Oncol. 1985 Jun;3(6):827-41. doi: 10.1200/JCO.1985.3.6.827. PMID 2409240
- [Background] Ruijter E, van de Kaa C, Miller G, Ruiter D, Debruyne F, Schalken J. Molecular genetics and epidemiology of prostate carcinoma. Endocr Rev. 1999 Feb;20(1):22-45. doi: 10.1210/edrv.20.1.0356. No abstract available. PMID 10047972
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2007-C-0100.html